CLINICAL TRIAL: NCT02584010
Title: Comparative, Open, Randomized Trial Between Two Silicon-based Products to Treat Postoperative Scars
Brief Title: Efficacy Study of Two Silicon-based Products to Treat Scars
Acronym: Kelofin
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: All-M-42361-01-08-14
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Scars
Keywords: Postoperative scars; Cicatrix; Cicatrization
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kelofin Aerosol (Experimental): Silicon-based Aerosol that will be applied over the postoperative scar two times a day
  Interventions: Other: Silicon-based aerosol
- Kelofin Gel (Experimental): Silicon-based Gel that will be applied over the postoperative scar two times a day
  Interventions: Other: Silicon-based gel
- Control (No Intervention): This group will not receive any intervention as a control group.

INTERVENTIONS:
Other: Silicon-based aerosol — Apply twice a day over the postoperative scar
  Other Names: Kelofin Aerosol
  Arms: Kelofin Aerosol
Other: Silicon-based gel — Apply twice a day over the postoperative scar
  Other Names: Kelofin Gel
  Arms: Kelofin Gel

SUMMARY:
This study aims to determine if a silicon-based gel and a silicon-based aerosol are effective in the treatment of postoperative scars.

DETAILED DESCRIPTION:
Improve the final aspect of scars, have been a challenge for medicine. Silicon based products have been used in various ways to prevent hypertrophic scars and keloids since 1980. A great percentage of studies shows that silicon-based products improves the aspect of scars in different pathologies. The main objective of this trial is to evaluate the efficacy, using the Vancouver scale, of two silicon-based products (Kelofin gel and Kelofin aerosol) after 180 days.

300 participants that meet all the inclusion criteria and are not classified in any of the exclusion criteria will be randomly allocated to one of thre treatment groups( Kelofin Gel, Kelofin Aerosol and no treatment) of the study.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin phototype I, II, III or IV
* Participant that has a recent surgical scar on remodeling phase (14 ± 7 days after surgery) from the following: breast plastic with inframammary incision (fold beneath the breast) or abdominoplasty, cesarean section, hysterectomy (removal of the uterus), oophorectomy (removal of ovaries), oophoroplasty (removal of nodules, cysts, etc. of the ovaries), salpingectomy (removal of the fallopian tubes), tubal ligation, exploratory laparotomy and ectopic pregnancy (pregnancy outside the uterus) (Pfannenstiel access road - transverse incision , below the navel and approximately one finger above the symphysis pubis).

Exclusion Criteria:

* Skin Pathology in the product application area;
* Diabetes;
* Immune impairment;
* Use of systemic corticosteroids or immunosuppressants;
* Skin diseases: vitiligo, psoriasis, lupus, atopic dermatitis;
* Background reaction to silicon-based products;
* Other illnesses or medications that may interfere directly in the study or endanger the health of the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of scars clinical improvement | 180 days
  The scars will be evaluated by the Vancouver scale since the baseline visit until 180 days after the end of the treatment.

SECONDARY OUTCOMES:
Evaluation of scars color improvement | 180 days
  The scars will be evaluated by the equipment Mexameter (Courage+Khazaka®) since the baseline visit until 180 days after the end of the treatment.
Evaluation of scars measurement improvement | 180 days
  The scars will be evaluated by the equipment Optical 3D Skin Measuring Device PRIMOS Compact 5.075, since the baseline visit until 180 days after the end of the treatment.
Participants satisfaction regarding the treatment | 180 days
  Assess the satisfaction of participants regarding the treatment on each visit using a questionnaire on improving the healing process
Adverse events occurrence | 180 days
  Adverse events will be evaluated since the baseline visit until 180 days after the end of the treatment.